CLINICAL TRIAL: NCT01989624
Title: PAncreatic Adenocarcinoma in Hospital
Acronym: APACH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD064-13
Record Dates: First submitted 2013-11-06; First posted 2013-11-21 (Estimated); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Pancreatic adenocarcinoma; diagnosis; treatment
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic Adenocarcinoma

SUMMARY:
Few data are currently available in the literature on pancreatic adenocarcinoma in France. About 8,000 new cases each year in France. The 5-year survival for all stages combined is <5%. This is the only digestive cancer in which mortality / incidence ratio is 98%.

Epidemiological characteristics at diagnosis, the impact on the survival of recent advances related to surgery, adjuvant chemotherapy and new standard forms of adjuvant chemotherapy (FOLFIRINOX) are mispriced in real life.

The development of new drugs and the development of Phase II and III require a better understanding of the state of this disease in the country.

The main objective is to describe the characteristics of the pancreatic adenocarcinoma at diagnosis in France and make an inventory of diagnostic practices and support.

ELIGIBILITY:
Inclusion Criteria:

* Living in France
* Pancreatic adenocarcinoma histologically or cytologically proven
* primary diagnosis
* Agreed to participate

Exclusion Criteria:

* Suspected pancreatic adenocarcinoma histologically or cytologically unproven
* Refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient in hepatogastroenterology in general hospital
Sampling Method: Non-Probability Sample
Enrollment: 1204 (Actual)
Dates: Start 2013-10-18 (Actual); Primary Completion 2015-12-04 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Survival | patient death (following during 5 year)

CONTACTS AND LOCATIONS:
Overall Officials: Roger FAROUX, PH, Principal Investigator — Centre hospitalier départemental Vendée
Locations (66):
- CH de Jolimont, Jolimont, Belgium
- France (65):
  - CH Gabriel Martin, Saint-Paul, La Réunion
  - CHIAP, Aix-en-Provence
  - CH Angoulême, Angoulême
  - CH d'Aubenas, Aubenas
  - CH Auch, Auch
  - CH Robert Ballanger, Aulnay-sous-Bois
  - CH Avignon, Avignon
  - CH Bagnols sur Ceze, Bagnols-sur-Cèze
  - CH Bayeux, Bayeux
  - CH Béziers, Béziers
  - CH Blois, Blois
  - CH Bourg en Bresse, Bourg-en-Bresse
  - CH de Bourges, Bourges
  - CH Nord Deux Sèvres, Bressuire
  - CH Saint Camille, Bry-sur-Marne
  - HPA Castres Mazamet, Castres
  - CH Chambery, Chambéry
  - CH Chartres, Chartres
  - CH Chalons en champagne, Châlons-en-Champagne
  - CH Haut Anjou, Château-Gontier
  - CH Châteauroux, Châteauroux
  - Ch Cholet, Cholet
  - CH Compiègne Noyon, Compiègne
  - CH sud francilien, Corbeil-Essonnes
  - CH de Creil, Creil
  - CHI Créteil, Créteil
  - CH Dourdan, Dourdan
  - CH Draguignan, Draguignan
  - CH Dreux, Dreux
  - CH Simone Veil, Eaubonne
  - CH Forcilles, Férolles
  - Chicas, Gap
  - CH Gonesse, Gonesse
  - Centre hospitalier départemental Vendée, La Roche-sur-Yon
  - Centre Hospitalier de Lagny, Lagny-sur-Marne
  - CH du Mans, Le Mans
  - Lens, Lens
  - Centre Hospitalier Côté de lumière, Les Sables-d'Olonne
  - Hôpital des chanaux, Mâcon
  - Centre Hospitalier de Meaux, Meaux
  - CH Melun, Melun
  - CHR de Mercy-Metz, Metz
  - CHAM, Montargis
  - CH Montauban, Montauban
  - Centre Hospitalier Montelimar, Montélimar
  - CH Montfermeil, Montfermeil
  - CH Niort, Niort
  - CHG Oloron, Oloron-Sainte-Marie
  - CHR Orléans, Orléans
  - CH François Mitterand, Pau
  - Centre Hospitalier de Perpignan, Perpignan
  - CHI Poissy Saint Germain, Poissy
  - CH Pontoise, Pontoise
  - CH de la région d'Annecy, Pringy
  - CH Quimper, Quimper
  - CH Roubaix, Roubaix
  - Centre hospitalier Yves Le Foll, Saint-Brieuc
  - CH de la Fontaine, Saint-Denis
  - CH Saint Quentin, Saint-Quentin
  - Centre Hospitalier de Bigorre, Tarbes
  - CH Sainte Musse, Toulon
  - CH Tourcoing, Tourcoing
  - CH Valenciennes, Valenciennes
  - CHBA de Vannes, Vannes
  - CHIV Villeneuve Saint-Georges, Villeneuve-Saint-Georges